CLINICAL TRIAL: NCT06059612
Title: Treatment of Upper Cluneal Nerve Entrapment Syndrome for Reduction of Low Back Pain: Single-arm Experimental Study
Brief Title: Treatment of Upper Cluneal Nerve Entrapment Syndrome for Reduction of Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLU-1
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Superior Cluneal Nerve Entrapment
Keywords: Superior cluneal nerve; nerve entrapment
MeSH Terms: conditions — Nerve Compression Syndromes | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Superior cluneal nerve entrapment (SCN) will be treated with local steroid injection
  Interventions: Procedure: injection

INTERVENTIONS:
Procedure: injection — steroid injection into superior cluneal nerve

SUMMARY:
Superior cluneal nerve entrapment (SCN) is a painful symptomatic condition related to compression by the thoracolumbar and gluteal bands of nerve outcrop, above the iliac crest. This syndrome is not considered in the classical differential diagnosis of lumbosacral spine disorders and is almost unknown in Italy.

It is a neuropathic pain, acute, subacute, or chronic, evoked by mechanical stress at the level of the sensory territory corresponding to the superior cluneal nerve, easily found anatomically and evoked at a trigger point on the posterior iliac crest approximately 70mm from the midline and 45mm from the posterior superior iliac spine.

SCN entrapment syndrome represents a not so infrequent syndrome. It is easily framed and treatment is effective in most cases. Therefore, diagnosis and treatment of this syndrome represents an excellent option in all those patients with low back pain that cannot be otherwise framed and resolved.

ELIGIBILITY:
Inclusion Criteria:

* patients with age between 18 and 99 years
* male and female sex
* superior cluneal nerve trigger point positivity at clinical evaluation
* absence of urgent criteria for spinal surgery

Exclusion Criteria:

* patients younger than 18 years old
* patients who have not given consent to be included in the study
* patients with negative upper cluneal nerve trigger point - emergency criteria for spine surgery
* pregnant women - patients allergic to local anesthetic
* patients with language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
numerical rating scale (NRS) | at baseline (day 0)
  NRS is a numerical scale for assessing pain exclusively. It is precisely a numerical scale ranging from 0 to 10 where the degree of pain perceived by the patient is expressed in an increasing manner. The value 0 corresponds to the 'absence of pain, the valor
numerical rating scale (NRS) | after 45 days
  NRS is a numerical scale for assessing pain exclusively. It is precisely a numerical scale ranging from 0 to 10 where the degree of pain perceived by the patient is expressed in an increasing manner. The value 0 corresponds to the 'absence of pain, the valor
Owestry Disability Index (ODI) | at baseline (day 0)
  The ODI score is a scorecard on daily activities and the degree of limitation experienced by the patient with low back pain.
  The form consists of 10 multiple-choice questions (5 options) regarding different aspects of daily life such as pain intensity, personal care, walking, climbing stairs, standing up, sleeping, sexual sphere, social sphere, and traveling. At the end of the assessment, a percentage is assigned where 100% expresses the absence of limitations in performing daily activities. The further away from the maximum threshold, the greater the degree of disability the patient experiences.
Owestry Disability Index (ODI) | after 45 days
  The ODI score is a scorecard on daily activities and the degree of limitation experienced by the patient with low back pain.
  The form consists of 10 multiple-choice questions (5 options) regarding different aspects of daily life such as pain intensity, personal care, walking, climbing stairs, standing up, sleeping, sexual sphere, social sphere, and traveling. At the end of the assessment, a percentage is assigned where 100% expresses the absence of limitations in performing daily activities. The further away from the maximum threshold, the greater the degree of disability the patient experiences.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuniya H, Aota Y, Kawai T, Kaneko K, Konno T, Saito T. Prospective study of superior cluneal nerve disorder as a potential cause of low back pain and leg symptoms. J Orthop Surg Res. 2014 Dec 31;9:139. doi: 10.1186/s13018-014-0139-7. PMID 25551470
- [Result] Morimoto D, Isu T, Kim K, Chiba Y, Iwamoto N, Isobe M, Morita A. Long-term Outcome of Surgical Treatment for Superior Cluneal Nerve Entrapment Neuropathy. Spine (Phila Pa 1976). 2017 May 15;42(10):783-788. doi: 10.1097/BRS.0000000000001913. PMID 27669049
- [Result] Bodner G, Platzgummer H, Meng S, Brugger PC, Gruber GM, Lieba-Samal D. Successful Identification and Assessment of the Superior Cluneal Nerves with High-Resolution Sonography. Pain Physician. 2016 Mar;19(3):197-202. PMID 27008294